CLINICAL TRIAL: NCT03223753
Title: A Randomized Web-Based Physical Activity Intervention Among Children and Adolescents With Cancer
Brief Title: Web-Based Physical Activity Intervention in Improving Long Term Health in Children and Adolescents With Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ALTE1631; NCI-2017-01219 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ALTE1631 (Other: Children's Oncology Group); COG-ALTE1631 (Other: DCP); ALTE1631 (Other: CTEP); R01CA193478 (NIH); UG1CA189955 (NIH)
Record Dates: First submitted 2017-07-11; First posted 2017-07-21 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Carcinoma In Situ; Hematopoietic and Lymphatic System Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Carcinoma in Situ | interventions — Early Intervention, Educational; Educational Status; Methods; Physical Examination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (tracking device, limited version of device) (Active Comparator): Patients receive educational handouts about physical activity and are encouraged to increase physical activity to at least 420 minutes per week. Patients wear physical activity tracking device daily and upload data at least once a week to the device app/website. Patients also access the limited version of device app/website to get basic information related to their physical activity for 6 months.
  Interventions: Other: Educational Intervention; Other: Internet-Based Intervention; Other: Laboratory Biomarker Analysis; Device: Medical Device Usage and Evaluation; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (tracking device, interactive-reward based device) (Experimental): Patients receive educational handouts about physical activity and are encouraged to increase physical activity to at least 420 minutes per week. Patients wear physical activity tracking device daily and upload data at least once a week to the device app/website. Patients also access the full version of the interactive-reward based device app/website to see their activity, earn activity points, see other's activity, and interact with other patients for 6 months.
  Interventions: Other: Educational Intervention; Other: Internet-Based Intervention; Other: Laboratory Biomarker Analysis; Device: Medical Device Usage and Evaluation; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Educational Intervention — Receive educational handouts about to physical activity
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
Other: Internet-Based Intervention — Access limited version of device app/website
  Arms: Arm I (tracking device, limited version of device)
Other: Internet-Based Intervention — Access full version of interactive reward-based device app/website
  Arms: Arm II (tracking device, interactive-reward based device)
Other: Laboratory Biomarker Analysis — Correlative studies
Device: Medical Device Usage and Evaluation — Wear physical activity tracking device
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized clinical phase III trial studies how well web-based physical activity intervention works in improving long term health in children and adolescents with cancer. Regular physical activity after receiving treatment for cancer may help to maintain a healthy weight and improve energy levels and overall health.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the effects of a rewards-and web-based physical activity intervention that includes structured social interaction between participants to the same web-based physical activity intervention that does not include structured social interaction on fitness among children and adolescents following treatment for cancer.

SECONDARY OBJECTIVES:

I. To evaluate the effect of a rewards-based, socially interactive web-based physical activity intervention on markers of cardiometabolic health among children and adolescents following treatment for cancer (compared to the same web-based physical activity intervention without social interaction).

II. To evaluate the effect of a rewards-based, socially interactive, web-based physical activity intervention on physical activity, quality of life, fatigue, and school attendance among children and adolescents following treatment for cancer (compared to the same web-based physical activity intervention without social interaction).

III. To determine if the effect of a rewards-based, socially interactive, web-based physical activity intervention on markers of cardiometabolic health is mediated by changes in fitness among children and adolescents following treatment for cancer (compared to the same web-based physical activity intervention without social interaction).

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive educational handouts about physical activity and are encouraged to increase physical activity to at least 420 minutes per week. Patients wear a physical activity tracking device daily and upload data at least once a week to the device app/website. Patients also access the limited version of the app/website to get basic information related to their physical activity. Patients will not be told of the details of earning of monetary incentives. Their activity will be monitored during the 6 month intervention period and will receive all earned gift cards or prizes after the intervention period ends. The patient will be encouraged to continue to wear the device for the remainder of the study, although they will no longer be earning monetary incentives.

ARM II: Patients receive educational handouts about physical activity and are encouraged to increase physical activity to at least 420 minutes per week. Patients wear a physical activity tracking device daily and upload data at least once a week to the device app/website. Patients also access the full version of the interactive-reward based device app/website to see their activity, earn activity points, see other's activity, and interact with other patients randomized to this study arm. Patients will receive additional details about how to earn gift cards or prizes for engaging in the intervention and will be rewarded for all earned incentives throughout the 6 month intervention period. The patient will be encouraged to continue to wear the device for the remainder of the study, although they will no longer be earning monetary incentives.

After completion of study, patients are followed up at 24 and 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* All cancer cases with an International Classification of Diseases for Oncology (ICD)-O histologic behavior code of two "2" (carcinoma in situ) or three "3" (malignant), in remission
* Patient must have completed curative therapy (surgery and/or radiation and/or chemotherapy) within the past 12 months at a Childrens Oncology Group (COG) institution
* Patients must have a performance status corresponding to Eastern Cooperative Oncology Group (ECOG) scores of 0, 1, or 2; use Lansky for patients =< 16 years of age
* At the time of consent, patient or parent/guardian reports less than 420 minutes of moderate to vigorous physical activity over the last week
* Patient and at least one parent/guardian are able to read and write English, Spanish, and/or French; at least 1 parent/guardian must be able to read and write English, Spanish, and/or French in order to assist the patient with using their physical activity tracking device account
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Exclusion Criteria:

* Patients with previous hematopoietic stem cell transplant (HSCT)
* Patients with significant concurrent disease, illness, psychiatric disorder or social issue that would compromise patient safety or compliance with protocol therapy, or interfere with consent, study participation, follow up, or interpretation of study results
* Female patients who are pregnant are not eligible; women of childbearing potential require a negative pregnancy test
* Female patient who is postmenarcheal and has not agreed to use an effective contraceptive method (including abstinence) for the duration of study participation
* Patients with a cognitive, motor, visual or auditory impairment that prevents computer use (e.g. unresolved posterior fossa syndrome) are not eligible

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Physiologic cost index (PCI) | Up to 24 weeks (end of intervention)
  Differences in PCI will be compared between groups at the end of the intervention. Intent to treat analysis of variance (either transforming the data or employing a non-parametric equivalent if the data are not normally distributed) controlling for the stratification factors (sex, age, and treatment related risk group) will be used for comparison. General linear mixed models will be utilized to evaluate the effects of group assignment on changes in PCI over time to account for repeated measures on individual children, and for potential random effects such as original treating institution.

SECONDARY OUTCOMES:
Change in markers of cardiometabolic health | Baseline up to 48 weeks post intervention
  Markers of Cardiometabolic health include blood pressure, body mass index, waist to height ration, fasting insulin, glucose, and lipid levels. Differences in these markers between randomized groups and the effects of group assignment on changes over time will be evaluated.
Change in inflammation | Baseline up to 48 weeks post intervention
  Markers of an Inflammatory state include High sensitivity C-reactive protein, interleukin-6, and tumor necrosis factor alpha. Differences in these markers between groups and the effects of group assignment on changes over time will be evaluated.
Change in quality of life | Baseline up to 48 weeks post intervention
  Will be assessed using Pediatric Quality of Life (PedsQL) 4.0 Generic Core Scale. The 23-item PedsQL Generic Core Scales were designed to measure the core dimensions of health as delineated by the World Health Organization, as well as role (school) functioning. Scores range from 0-100, higher is better. There are four scales (Physical Functioning, Emotional Functioning, Social Functioning, and School Functioning). Emotional, Social and School Functioning can be combined to create a psychosocial summary (summed and divided by total number of items). Differences between groups and the effects of group assignment on changes over time will be evaluated.
Change in fatigue | Baseline up to 48 weeks post intervention
  Will be assessed using Pediatric Quality of Life Multidimensional Fatigue Scale. The PedsQL Multidimensional Fatigue Scale was designed as a generic symptom-specific instrument to measure fatigue in patients with acute and chronic health conditions as well as healthy school and community populations. It has three dimensions, general fatigue, sleep/rest fatigue and cognitive fatigue. Scores range from 0-100 and items are summed and divided by the total to get the mean. Differences between groups and the effects of group assignment on changes over time will be evaluated.
Change in school attendance | Baseline up to 48 weeks post intervention
  Will be assessed using parent report. Differences between groups and the effects of group assignment on changes over time will be evaluated.
Markers of cardiometabolic health | Up to 48 weeks post intervention
  Markers of cardiometabolic health include blood pressure, body mass index, waist to height ration, fasting insulin, glucose, and lipid levels. It will be determined if the effect of an interactive web-based physical activity intervention on markers of cardiometabolic health is mediated by changes in fitness among children and adolescents following treatment for acute lymphoblastic leukemia. A causal inference approach will evaluate whether group assignment results in an improved outcome in the presence of a lower PCI. This requires decomposing the averaged total effect into indirect and direct effects of group assignment of on the cardiometabolic outcomes. A principal stratification method will be used that classifies participants into strata based on their performance on the PCI (mediator variable) for each group of the randomized intervention. Mediation analyses would then be based on intent-to-treat effects of group assignment on cardiometabolic health outcome within each strata.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten K Ness, Principal Investigator — Children's Oncology Group
Locations (118):
- United States (113):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Banner Children's at Desert, Mesa, Arizona
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - Palms West Radiation Therapy, Loxahatchee Groves, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Tampa General Hospital, Tampa, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Atrium Health Navicent, Macon, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Advocate Children's Hospital-Park Ridge, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Tufts Children's Hospital, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Missouri Children's Hospital, Columbia, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Sciences Center-Amarillo, Amarillo, Texas
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - UMC Cancer Center / UMC Health System, Lubbock, Texas
  - Vannie Cook Children's Clinic, McAllen, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Carilion Children's, Roanoke, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
- Canada (5):
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Child Health Centre, St. John's, Newfoundland and Labrador
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario

REFERENCES:
- [Derived] Ware ME, Kadan-Lottick NS, Devidas M, Terrell S, Chow EJ, Ehrhardt MJ, Hardy KK, Chemaitilly W, Hein W, Winick N, Teachey D, Esbenshade A, Armenian SH, Partin RE, Ness KK. Design and methods of a randomized web-based physical activity intervention among children with cancer: A report from the Children's Oncology Group. Contemp Clin Trials. 2022 Nov;122:106961. doi: 10.1016/j.cct.2022.106961. Epub 2022 Oct 10. PMID 36228982